CLINICAL TRIAL: NCT05815160
Title: A Phase 1 Dose-Escalation and Expansion Study to Assess Safety and Preliminary Antitumor Activity of Debio 0123 in Combination With Carboplatin and Etoposide in Adult Participants With Small Cell Lung Cancer That Recurred or Progressed After Previous Standard Platinum-Based Therapy
Brief Title: Debio 0123 in Combination With Carboplatin and Etoposide in Adult Participants With Small Cell Lung Cancer That Recurred or Progressed After Previous Standard Platinum-Based Therapy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Debio 0123-SCLC-104; 2024-510980-40-00 (EU CTIS Number); U1111-1302-8787 (Other: WHO Unique Trial identifier)
Record Dates: First submitted 2023-03-09; First posted 2023-04-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Small Cell Lung Cancer Recurrent
Keywords: Small cell lung cancer (SCLC); Recurrent; Debio 0123; Carboplatin; Etoposide; WEE1 inhibitor; WEE-1 inhibitor; Platinum-based therapy; Platinum-based chemotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma; Recurrence | interventions — Etoposide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation: Debio 0123 + Etoposide + Carboplatin (Experimental): Participants will receive Debio 0123 escalating doses, orally along with etoposide IV infusion and carboplatin IV infusion in 21-day cycles until disease progression or death or end of study.
  Interventions: Drug: Debio 0123; Drug: Etoposide; Drug: Carboplatin
- Part 2: Dose Expansion: Debio 0123 + Etoposide + Carboplatin (Experimental): Participants will receive Debio 0123 recommended dose determined in Part 1 of the study, orally along with etoposide IV infusion and carboplatin IV infusion in 21-day cycles until disease progression or death or end of study.
  Interventions: Drug: Debio 0123; Drug: Etoposide; Drug: Carboplatin

INTERVENTIONS:
Drug: Debio 0123 — Administered as capsules.
Drug: Etoposide — Administered as IV infusion.
Drug: Carboplatin — Administered as IV infusion.

SUMMARY:
The primary purpose of part 1 (dose escalation) of this study is to identify the recommended dose and to characterize the safety and tolerability of Debio 0123 in combination with carboplatin and etoposide.

The primary purpose of part 2 (dose expansion) of this study is to characterize the safety and tolerability of Debio 0123 at the recommended dose when administered in combination with carboplatin and etoposide.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed SCLC
2. Tumor that is not bleeding
3. Prior platinum-based chemotherapy (carboplatin and/or cisplatin)

   * Part 1 (dose escalation): Recurrence or progression after a minimum of 45 days since the last dose of prior standard platinum-based therapy
   * Part 2 (expansion): Recurrence or progression after a minimum of 90 days since the last dose of prior standard platinum-based therapy
4. Measurable disease per RECIST 1.1
5. Willingness and ability to undergo tumor biopsy unless an archived tumor sample is available
6. ECOG performance status of 0-1
7. Life expectancy of at least 3 months in the best judgment of the Investigator
8. Adequate bone marrow, hepatic and renal function, adequate coagulation status
9. Willingness and ability to comply with scheduled visits, study treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Use of an investigational agent or medical device within 28 days prior to first dose of study treatment.
2. History of other malignancies requiring active treatment in the last 2 years prior to first dose of study treatment, except for superficial bladder cancers, ductal carcinoma in situ or other carcinomas in situ, and non-melanoma skin cancers (basal cell/squamous cell skin cancer) that have been treated with curative intent.
3. History of myocardial infarction or stroke in the last 6 months prior to first dose of study treatment, congestive heart failure greater than New York Heart Association (NYHA) class II, unstable angina pectoris, unexplained recurrent syncope, cardiac arrhythmia requiring treatment, known family history of sudden death from cardiac-related causes before the age of 50, or any cardiotoxicity experienced after previous chemotherapy.
4. Left ventricular ejection fraction (LVEF) below 55%.
5. QTcF >450 ms, history of congenital long QT syndrome, or clinically significant conduction abnormality, or any conduction abnormality that may increase the risk of TdP.
6. Clinically significant gastrointestinal abnormality that could affect the absorption of orally administered drugs
7. Major surgery ≤4 weeks prior to first dose of study treatment or incomplete recovery from the surgical procedure at the time of the first dose of study treatment.
8. Radiographic findings showing tumor involvement with large blood vessels or poor demarcation from them with increased risk for bleeding.
9. Radiographic findings of Interstitial lung disease (ILD) that are considered clinically significant.
10. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
11. Any infection requiring the systemic use of an antibiotic or antiviral agent.
12. Known Hepatitis C virus (HCV), Hepatitis B virus (HBV), or Human Immunodeficiency Virus (HIV) infection. Participants with past infections that have been cured may be enrolled.
13. Immunization with live or live-attenuated vaccine within 28 days prior to first dose of study treatment.
14. Inability or unwillingness to swallow oral medications.
15. Anticancer treatment (including chemotherapy), monoclonal antibodies/biologics, or radiotherapy with curative intent within 28 days prior to first dose of study treatment. Palliative radiation is allowed up to 1 week prior to study treatment start.
16. Unresolved AEs or toxicities due to previous treatments >Grade 1. Note: Participants with ≤Grade 2 alopecia or endocrinopathies controlled by replacement therapy are exceptions and may qualify for the study.
17. Hypersensitivity to Debio 0123, etoposide or carboplatin, or any of the excipients found in the formulations for Debio 0123, etoposide, or carboplatin. If a prior hypersensitivity to carboplatin has been observed but a successful desensitization was performed for the participant, he or she may be eligible for the study.
18. Prior exposure to any WEE1 inhibitor

Note: Other inclusion/exclusion criteria mentioned in the protocol may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants Experiencing Dose-limiting Toxicities (DLTs) | Cycle 1 (Cycle=21 days)
Parts 1 and 2: Number of Participants With at Least One Treatment Emergent Adverse Event (TEAE) | Approximately up to 44 months
Parts 1 and 2: Number of Participants With Clinically Significant Abnormalities in Laboratory, Vital Signs, Electrocardiogram (ECG), and Echocardiogram Parameters | Approximately up to 44 months
Parts 1 and 2: Change From Baseline in Eastern Cooperative Oncology Group Performance Status (ECOG PS) | Baseline up to approximately 44 months

SECONDARY OUTCOMES:
Parts 1 and 2: Trough Concentration (Ctrough) of Debio 0123 and its Metabolite | For Part 1: Predose from Day 2 to Day 11 of Cycle 1; For Part 2: Predose from Day 3 to Day 10 of Cycle 1 and only Day 8 of subsequent cycles up to Cycle 5 (Cycle=21 days)
Parts 1 and 2: Maximum Plasma Concentration (Cmax) of Debio 0123 and its Metabolite | For Part 1: Multiple timepoints post dose from Day 1 to Day 11 of Cycle 1 (Cycle=21 days); For Part 2: Will be derived from the population Pharmacokinetic (PK) model using the sparse samples collected
Parts 1 and 2: Area Under the Concentration Curve Over 24 hours (AUC24h) of Debio 0123 and its Metabolite | For Part 1: Multiple timepoints post dose from Day 1 to Day 11 of Cycle 1 (Cycle=21 days); For Part 2: Will be derived from the population PK model using the sparse samples collected
Part 1: Time to Maximum Plasma Concentration (tmax) of Debio 0123 and its Metabolite | Multiple timepoints post dose from Day 1 to Day 11 of Cycle 1 (Cycle=21 days)
Part 1: Area Under the Concentration Curve up to the Last Measurable Concentration (AUClast) of Debio 0123 and its Metabolite | Multiple timepoints post dose from Day 1 to Day 21 of Cycle 1 and Day 1 of Cycle 2 (Cycle=21 days)
Part 1: Area Under the Concentration Curve up to Infinity (AUCinf) of Debio 0123 and its Metabolite | Multiple timepoints post dose from Day 1 to Day 21 of Cycle 1 and Day 1 of Cycle 2 (Cycle=21 days)
Part 1: Apparent Terminal Half-life (t1/2) of Debio 0123 and its Metabolite | Multiple timepoints post dose from Day 1 to Day 21 of Cycle 1 and Day 1 of Cycle 2 (Cycle=21 days)
Part 1: Apparent Clearance (CL/F) of Debio 0123 | Multiple timepoints post dose from Day 1 to Day 21 of Cycle 1 and Day 1 of Cycle 2 (Cycle=21 days)
Part 1: Apparent Volume of Distribution (Vd/F) of Debio 0123 | Multiple timepoints post dose from Day 1 to Day 21 of Cycle 1 and Day 1 of Cycle 2 (Cycle=21 days)
Part 1: Maximum Plasma Concentration (Cmax) of Etoposide | Multiple timepoints from administration to post dose from Day 1 to Day 3 of Cycle 1 (Cycle=21 days)]
Part 1: Area Under the Concentration Curve Over 24 hours (AUC24h) of Etoposide | Multiple timepoints post dose from Day 1 to Day 5 of Cycle 1 (Cycle=21 days)
Part 1: Trough Concentration (Ctrough) of Etoposide | Predose from Day 2 to Day 5 of Cycle 1 (Cycle=21 days)
Part 1: Maximum Plasma Concentration (Cmax) of Carboplatin | Multiple timepoints from administration up to 6 hours post dose on Day 1 of Cycle 1 (Cycle=21 days)
Parts 1 and 2: Percentage of Participants With Best Overall Response (BOR) Assessed as per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 Criteria | From the start of study treatment until disease progression or end of study (up to approximately 44 months)
Parts 1 and 2: Percentage of Participants With Objective Response (OR) Assessed as per RECIST 1.1 Criteria | Up to end of study (approximately 44 months)
Parts 1 and 2: Percentage of Participants With Disease Control (DC) Assessed as per RECIST 1.1 Criteria | From the start of study treatment until disease progression or end of study (up to approximately 44 months)
Parts 1 and 2: Duration of Response (DOR) Assessed as per RECIST 1.1 Criteria | Up to disease progression or end of study (approximately 44 months)
Parts 1 and 2: Progression Free Survival (PFS) Assessed as per RECIST 1.1 Criteria | From the start of study treatment until disease progression or death or end of study (up to approximately 44 months)
Part 2: Overall Survival | From the start of study treatment until death from any cause or end of study (up to approximately 44 months

CONTACTS AND LOCATIONS:
Locations (13):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
- Spain (11):
  - Hospital Universitario de A Coruna, A Coruña
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Institut Catala D'Oncologia - Badalona, Barcelona
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro. START Madrid - Centro Integral Oncológico Clara Campal (CIOCC), Madrid
  - NEXT Oncology Madrid, Madrid
  - Hospital Quironsalud Malaga, Málaga
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No